CLINICAL TRIAL: NCT03321799
Title: Comparison of Negative Pressure Wound Therapy Versus Conventional Dressings for the Prevention of Wound Complications Following Revision Total Hip Arthroplasty: A Prospective, Randomized, Controlled Trial
Brief Title: Comparison of Negative Pressure Wound Therapy vs. Conventional Dressings for Prevention of Wound Complications After Revision THA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16111608
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Infection, Drainage
MeSH Terms: conditions — Infections | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sterile Antimicrobial Dressings (Active Comparator): Control group, current hospital standard. AQUACEL is left in place for 7 days unless it becomes saturated over 50%, which requires a premature dressing change.
  Interventions: Device: Sterile Antimicrobial Dressings
- Negative pressure wound therapy (NPWT) (Experimental): Experimental group. Negative pressure wound therapy bandage applied intra-operatively by a physician on the treatment team.
  The dressing will be removed after 7 days postoperatively, or if the battery power stops earlier.
  Interventions: Device: Negative Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Device: Negative Pressure Wound Therapy (NPWT) — A computer randomization system will be used on the day of surgery to allocate patients to either the conventional or NPWT dressing. Due to the nature of this study, blinding of patients and surgeons to their allocated cohort will not be possible.
  Arms: Negative pressure wound therapy (NPWT)
Device: Sterile Antimicrobial Dressings — Control group, current hospital standard.
  Arms: Sterile Antimicrobial Dressings

SUMMARY:
Wound complications and surgical site infections following revision total joint arthroplasty result in significant morbidity and cost. To the investigators knowledge, no prospective, randomized controlled trials have examined the rate of wound complications, infection, and reoperation following revision total hip arthroplasty when treated with negative pressure wound therapy (NPWT) versus sterile dressings. The investigators hypothesize that the rate of wound complications, infections, and subsequent procedures in patients undergoing revision THA treatment will demonstrate a statistically and clinically relevant decrease when using NPWT versus sterile dressing.

DETAILED DESCRIPTION:
Wound complications and surgical site infections (SSI) following revision total joint arthroplasty result in significant morbidity and cost. Persistent incisional drainage following total joint arthroplasty (TJA) has been reported to occur in 1% to 3% of patients. Drainage persisting greater than 48 hours has been reported as a risk factor for the development of an acute periprosthetic joint infection (PJI), with each additional day of wound drainage increasing the infection risk by 29-42%. Consequently, continued wound drainage has been shown to potentially increase the economic burden through longer hospital stays and subsequent surgical procedures. To the investigators knowledge, no prospective, randomized controlled trials have examined the rate of wound complications, infection, and reoperation following revision total hip arthroplasty when treated with NPWT versus sterile dressings. The investigators hypothesize that the rate of wound complications, infections, and subsequent procedures in patients undergoing revision THA treatment will demonstrate a statistically and clinically relevant decrease when using NPWT versus sterile dressing. The investigators will utilize a prospective, randomized, controlled study design to assess the efficacy of negative pressure wound therapy (NPWT) on the rate of wound complications, surgical site infections (SSIs), and reoperations after revision total hip arthroplasty (THA). For 90 days after surgery, the wound complications, including wound dehiscence, prolonged drainage for >7 days postoperatively, hematoma formation, surgical site infection, or periprosthetic joint infection that requires postoperative interventions, and reoperation will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age undergoing a revision total hip arthroplasty procedure to include:
* Conversion of a prior open hip surgery (i.e. open reduction internal fixation of a proximal femur fracture) to a total hip arthroplasty
* Aseptic revision for a diagnosis of component loosening, osteolysis, or revision procedure for periprosthetic fracture that requires revision of a component of the THA prosthesis (excluded isolated open reduction internal fixation of the fracture or initial placement of a hemi- or total hip arthroplasty)
* Septic revision surgery including irrigation and debridement of a postoperative infection or hematoma, one-stage exchange for acute postoperative infection, explantation and placement of an antibiotic cement spacer
* Reimplantation of a THA following placement of an antibiotic-loaded cement spacer
* The incision can be closed primarily without muscle flaps or skin grafting
* Willingness to undergo randomization and return for all scheduled visits

Exclusion Criteria:

* Patients requiring a muscle flap or skin grafting for wound closure
* Pregnant or lactating female
* Known sensitivity to the study product components (adhesives, etc.)
* Allergy to silver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Wound complications | 90 days
  Wound complications within 90 days of a revision total hip arthroplasty include: wound dehiscence, prolonged drainage for >7 days postoperatively, hematoma formation, surgical site infection, or periprosthetic joint infection that requires postoperative interventions (i.e. unplanned office visits, topical application of antibiotics or PO antibiotics, in-office wound debridement or removal of suture material, hematoma aspiration and drainage) or a return to the operating room/reoperation.

SECONDARY OUTCOMES:
Reoperation | 90 days
  Reoperation for a wound complication, surgical site infection, or periprosthetic joint infection within 90 days of the revision THA
Cost comparison | 90 days
  Cost comparison between the NPWT and routine dressing changes within 90 days to include the potential costs of postoperative interventions and reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Denis Nam, MD, MSc, Principal Investigator — Rush University Medical Center
Locations (1):
- Anne DeBenedetti, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently there is no plan to share IPD and if that is decided in the future, that information will be de-identified and in compliant with HIPAA regulations